CLINICAL TRIAL: NCT00563173
Title: A Phase I/IIa Open-Label, Dose Ranging, Parallel, Safety, Tolerability and Efficacy Study of i.m. Administered CHRONVAC-C® in Combination With Electroporation in Chronic HCV Genotype 1 Infected and Treatment Naïve Patients With Low Viral Load
Brief Title: Phase I/IIa Dose Ranging CHRONVAC-C® Study in Chronic HCV Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tripep AB (Industry)
Collaborators: Inovio Pharmaceuticals (Industry)
Responsible Party: Prof. Anders Vahlne/CEO, Tripep AB
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVC-201; EudraCT No. 2007-002901-33
Record Dates: First submitted 2007-11-23; First posted 2007-11-26 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Hepatitis C Virus Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Other): Low dose
  Interventions: Drug: CHRONVAC-C®
- 2 (Other): Medium dose
  Interventions: Drug: CHRONVAC-C®
- 3 (Other): High dose
  Interventions: Drug: CHRONVAC-C®

INTERVENTIONS:
Drug: CHRONVAC-C® — DNA vaccine, solution for injection, i.m. administration in combination with electroporation

SUMMARY:
The purpose of this study is to evaluate if the DNA vaccine CHRONVAC-C® intended for future treatment of Hepatitis C infections is safe and tolerated when administered to HCV infected individuals with a low viral load. In addition the capability of the vaccine to induce an immune response and the effect on viral load will be studied. In order to increase the uptake of the vaccine the intra muscular injection is combined with electroporation, meaning that a brief electric field is applied to the injection site resulting in temporary pores in the cell membranes that allows the vaccine to enter the cells.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient 18 -65 years of age with a known chronic hepatitis C infection.
* Genotype 1 infection.
* Viral load equal to or less than 800.000 IU/mL.
* BMI less than 30.
* Considered probable that the deltoid muscles (left and right) of the patient will be reached at vaccination using a 12.7 mm cannula for injection and a 15 mm applicator tip for electroporation.
* Written informed consent obtained, and a copy provided to the patient.
* Patient legally competent and able to communicate effectively with the study personnel.
* Patient likely to co-operate and attend the clinic at the appointed times during the study.

Exclusion Criteria:

* Patient having clinically significant concomitant diseases other than HCV in the medical history to the discretion of the investigator.
* Patient having clinically significant findings on physical examination, vital signs, ECG or clinical laboratory evaluations to the discretion of the investigator.
* Patient having clinical or biochemical signs of cirrhosis.
* Positive hepatitis B surface antigen (HBsAg).
* Positive HIV antigen or antibody test.
* Patient having an ongoing and/or known viral infection other than HCV that requires treatment and/or special medical intention.
* Patient having received previous treatment for HCV.
* Radiation therapy or cytotoxic chemotherapeutic agents within 4 weeks prior to the first dose of study drug.
* Treatment with immunomodulating agents such as systemic corticosteroids, IL-2, IFN-alpha, IFN-beta, IFN-gamma within 4 weeks prior to the first dose of study drug.
* Treatment with NSAID within 10 days of the first dose of study drug.
* Immunization within 30 days of the first dose of the study drug.
* Patient having received an investigational drug product, or been enrolled in other investigational drug protocols within a period of 30 days prior to receiving the first dose of the study drug.
* Prior treatment with DNA therapy.
* Known allergy towards vaccines.
* Known abuse of alcohol, drugs or pharmaceuticals.
* History, signs or symptoms of a cardiac disease.
* Presence of an implantable pacemaker.
* Any metal implants within the treatment areas (close to the right and/or left deltoid muscles).
* Diagnoses of a serious psychiatric illness which may influence study participation.
* Female patient who is breast feeding.
* Female patient not clinically sterile (hysterectomy, tubal ligation or postmenopausal (amenorrhea > 1 year and FSH > 30 mU/ml) OR if not clinically sterile unwilling to use a reliable contraception method.
* Patient with a positive urine pregnancy test.
* Male patient unwilling to use condom for active prevention of pregnancy from first vaccination to 4 months after last injection.
* Patient or their immediate families being an investigator or site personnel directly affiliated with this study. Immediate family is defined as a spouse, parent, child or sibling, whether biologically or legally adopted.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of electroporation mediated i.m. delivery of CHRONVAC-C® in chronically HCV infected, treatment naive patients with low viral load. | From start of treatment to 24 weeks post treatment

SECONDARY OUTCOMES:
To provide information regarding dose related anti-viral immune response and dose related effect on viral load. | From start of treatment to 24 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ola RH Weiland, Professor, Principal Investigator — I73 Department of Infectious Diseases, Karolinska Institute, Karolinska University Hospital, Huddinge, Sweden; Anders Vahlne, Professor, Study Chair — Tripep AB; Matti Sällberg, Professor, Study Director — Tripep AB
Locations (2):
- Sweden (2):
  - I73 Department of Infectious Diseases, Karolinska Institute, Karolinska University Hospital, Huddinge, Stockholm
  - Department of Gastroenterology and Hepatology, Karolinska University Hospital, Solna, Stockholm